CLINICAL TRIAL: NCT05899296
Title: Assessment of Pain, Anxiety and Efficiency of NumBee Compared to Traditional Local Anesthetic Syringe (A Randomized Clinical Trial)
Brief Title: Assessment of Pain, Anxiety and Efficiency of NumBee Compared to Traditional Local Anesthetic Syringe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duaa Kamal Naji (Other)
Responsible Party: Sponsor-Investigator, Duaa Kamal Naji, Bachelor of dental surgery, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 576322
Record Dates: First submitted 2023-05-08; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Dental Phobia; Dental Anxiety; Anesthesia, Local; Needle Phobia
Keywords: Dental anxiety; Pain perception; Anesthetic efficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional syringe (Active Comparator): Dental anesthesia delivered by a traditional syringe
  Interventions: Device: Traditional dental syringe
- NumBee (Experimental): Dental anesthesia delivered by a novel needle-less syringe
  Interventions: Device: dental syringe ( NumBee)

INTERVENTIONS:
Device: dental syringe ( NumBee) — assess the capability of NumBee to reduce anxiety and pain during injection
  Arms: NumBee
Device: Traditional dental syringe — compare the level of anxiety of the traditional dental syringe and the Number dental syringe
  Arms: Traditional syringe

SUMMARY:
The study was conducted among a group of dental patients aged (6-8 years old) of both genders to assess the following variables in the needleless interparliamentary anesthesia (NUMBEE) compared to traditional local anesthesia:

1. Pain perception.
2. Pain related behaviors.
3. Dental anxiety
4. Anesthetic efficiency.
5. Patient acceptance and preference

DETAILED DESCRIPTION:
The prevalent phobia of needles and the associated rise in dental anxiety when using the traditional needle method of LA infiltration, the development of needle-free alternatives for local anesthetics became an urgent necessity. The NumBee (BioDent, Simi Valley, CA) is a new gadget that promises less pain administration of local anesthetic without the use of a hypodermic needle. It is a tiny metal cannula with a silicone-like covering that is used for intraligmentary injection without penetrating the periodontal ligament. This study was performed due to the lack of sufficient research on NumBee and since it meets a number of exceptional criteria, including being able to anesthetize just one tooth without having to do so for the entire alveolar dental nerve and having a needleless design that may be more appealing to children than the distressing appearance of traditional dental syringes.

ELIGIBILITY:
Inclusion Criteria:1. Patients with American Society of Anesthesiologists-1(ASA 1) health status (A completely healthy fit patient).

2. Not mentally retarded patient. 3. Cooperative patient, as determined by a behavioral rating of "positive" or "definitely positive" according to the Frankle behavior classification scale.

4. Without a history of dental visits.

-

Exclusion Criteria:

* 1. Mentally and medically compromised child. 2. Patient on medication that effect on the pain perception. 3. History of allergy to L.A.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
pain perception | five months
  checking the efficacy of NumBee syringe in reducing pain and anxiety in dental treatment

CONTACTS AND LOCATIONS:
Overall Officials: Duaa K Naji, Principal Investigator — University of Baghdad
Locations (1):
- University of Baghdad, Baghdad, KHARkh, Iraq

IPD SHARING:
Plan to Share IPD: Yes
it will be my pleasure to share and information with other resaercher
Supporting Information: Study Protocol
Time Frame: it will be available in 2023/2024 and for no limits
Access Criteria: data will be sent in e-mail for anyone wishes to access.
  Doaa.Kamal1202a@codental.uobaghdad.edu.iq